CLINICAL TRIAL: NCT02135107
Title: A Double-blind Comparative Study of the Efficacy and Safety of E3810 10mg Once and Twice Daily in Maintenance Therapy for PPI Resistant Gastroesophageal Reflux Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-J081-311
Record Dates: First submitted 2014-03-24; First posted 2014-05-09 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2018-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental)
  Interventions: Drug: Rabeprazole
- Arm B (Experimental)
  Interventions: Drug: Rabeprazole
- Arm C (Experimental)
  Interventions: Drug: Rabeprazole
- Arm D (Experimental)
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole 10 mg was administered orally twice daily during the treatment period for 8 weeks (unblinded).
  Other Names: E3810
  Arms: Arm A
Drug: Rabeprazole — Rabeprazole 20 mg was administered orally twice daily during the treatment period for 8 weeks (unblinded).
  Other Names: E3810
  Arms: Arm B
Drug: Rabeprazole — Rabeprazole 10 mg or 20 mg were administered orally twice daily during the treatment period (unblinded), and 10 mg was administered once daily during the maintenance period (double-blind).
  Other Names: E3810
  Arms: Arm C
Drug: Rabeprazole — Rabeprazole 10 or 20 mg were administered orally twice daily during the treatment period (unblinded), and 10 mg was administered twice daily during the maintenance period (double-blind).
  Other Names: E3810
  Arms: Arm D

SUMMARY:
The purpose of this study is to assess the efficacy and safety of rabeprazole 10mg once and twice daily in maintenance therapy for PPI resistant gastroesophageal reflux disease patients.

DETAILED DESCRIPTION:
This is randomized, multicenter, parallel-group, double-blind trial that investigates the efficacy and safety of rabeprazole 10mg twice daily over a period of 52 weeks. The 8-week Treatment Period (unblinded) was followed by a 52-week Maintenance Period (blinded). Participants with cure (modified Los Angeles Classification Grade N or Grade M) at the final endoscopy of the Treatment Period were entered into the Maintenance Period. Participants without cure were discontinued from the study. The participants in the Treatment Period were randomized to take Arm C or Arm D at a ratio of 1:1. The non-recurrence rate as endoscopically confirmed at 52 weeks shall be the primary end point, and this shall be examined through a randomized, multicenter, parallel-group, double-blind trial that investigates the efficacy and safety of rabeprazole 10mg twice daily over a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling all of the below criteria shall be eligible for the study:

1. Patients diagnosed with gastroesophageal reflux disease who are shown through endoscopic examination to have mucosal lesions (erosions, ulcers)
2. Patients shown through endoscopy not to have recovered despite administration of PPI once daily for eight weeks.
3. Patients over 20 years of age who have freely given their informed consent in writing to participation in the study.
4. Patients who, having received a full explanation of the matters that must be adhered to during the study, intend to adhere to their requirements, and are capable of doing so.

Exclusion Criteria:

Subjects fulfilling any of the following criteria shall be excluded from the study:

1. Patients considered candidates for surgical treatment of the upper gastrointestinal tract due to perforation, esophageal stricture, pyloric stenosis, esophageal varices, etc.
2. Patients with Zollinger-Ellison syndrome.
3. Patients with gastrointestinal hemorrhage.
4. Patients with serious cardiovascular disease, cerebrovascular disease, hematological disorders, renal disease, liver disease, malignant tumors, etc.
5. Patients with long segment Barrett's esophagus.
6. Patients with open gastric or duodenal ulcers.
7. Patients with drug allergies or a past history of drug allergies to PPI.
8. Patients who are taking other drugs under development, or have done so within 12 weeks prior to enrollment.
9. Patients who are, or may be pregnant, patients who wish to become pregnant during the study period, patients who are breastfeeding, and patients or their partners who do not wish to use reliable contraceptive measures.
10. Patients with a history of dependence on or abuse of drugs or alcohol within the past two years.
11. Other patients deemed unsuitable for inclusion in the study by the principal investigator or sub-investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- Japan (61):
  - Nagoya, Aichi-ken
  - Inzai, Chiba
  - Kamagaya, Chiba
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kōriyama, Fukushima
  - Annaka, Gunma
  - Fukuyama, Hiroshima
  - Asahikawa, Hokkaido
  - Ishikari, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Furukawa, Ibaraki
  - Tsuchiura, Ibaraki
  - Takamatsu, Kagawa-ken
  - Ichikikushikino-shi, Kagoshima-ken
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Suwa, Nagano
  - Beppu, Oita Prefecture
  - Fujiidera, Osaka
  - Hirakata, Osaka
  - Kishiwada, Osaka
  - Takatsuki, Osaka
  - Karatsu, Saga-ken
  - Ureshino, Saga-ken
  - Ageo, Saitama
  - Hiki, Saitama
  - Toda, Saitama
  - Wako, Saitama
  - Izumo, Shimane
  - Fujieda, Shizuoka
  - Hamamatsu, Shizuoka
  - Ōtawara, Tochigi
  - Adachi City, Tokyo
  - Bunkyo, Tokyo
  - Chūō, Tokyo
  - Koto, Tokyo
  - Minato, Tokyo
  - Nerima City, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Toshima City, Tokyo
  - Akita
  - Fukuoka
  - Hiroshima
  - Kochi
  - Kyoto
  - Nagasaki
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Yamagata

REFERENCES:
- [Derived] Kinoshita Y, Kato M, Fujishiro M, Masuyama H, Nakata R, Abe H, Kumagai S, Fukushima Y, Okubo Y, Hojo S, Kusano M. Efficacy and safety of twice-daily rabeprazole maintenance therapy for patients with reflux esophagitis refractory to standard once-daily proton pump inhibitor: the Japan-based EXTEND study. J Gastroenterol. 2018 Jul;53(7):834-844. doi: 10.1007/s00535-017-1417-z. Epub 2017 Nov 29. PMID 29188387

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabeprazole: 10 mg Twice Daily: Rabeprazole (10 mg) was administered orally twice daily during the treatment period for 8 weeks (unblinded).
- Rabeprazole: 20 mg Twice Daily: Rabeprazole (20 mg) was administered orally twice daily during the treatment period for 8 weeks (unblinded).
- Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily: Rabeprazole 10 mg or 20 mg was administered orally twice daily during the treatment period (unblinded), and 10 mg was administered once daily during the maintenance period (double-blind).
- Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily: Rabeprazole 10 mg or 20 mg was administered orally twice daily during the treatment period (unblinded), and 10 mg was administered twice daily during the maintenance period (double-blind).
Period: Treatment Period
Arm/Group | Rabeprazole: 10 mg Twice Daily | Rabeprazole: 20 mg Twice Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Started | 437 | 80 | 0 | 0
Completed | 305 | 54 | 0 | 0
Not Completed | 132 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Other | 115 | 24 | 0 | 0
Period: Maintenance Therapy Period
Arm/Group | Rabeprazole: 10 mg Twice Daily | Rabeprazole: 20 mg Twice Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Started | 0 (Treatment Phase only) | 0 (Treatment Phase only) | 178 (Only eligible participants entered into the Maintenance Therapy Period) | 181 (Only eligible participants entered into the Maintenance Therapy Period)
Completed | 0 | 0 | 163 | 161
Not Completed | 0 | 0 | 15 | 20
Not completed — Adverse Event | 0 | 0 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 4
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Rabeprazole: 10 mg Twice Daily: Rabeprazole 10 mg was administered orally twice daily during the treatment period for 8 weeks (unblinded).
- Rabeprazole: 20 mg Twice Daily: Rabeprazole 20 mg was administered orally twice daily during the treatment period for 8 weeks (unblinded).
- Total: Total of all reporting groups
Arm/Group | Rabeprazole: 10 mg Twice Daily | Rabeprazole: 20 mg Twice Daily | Total
Number analyzed (Participants) | 437 | 80 | 517
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (13.1) | 70.2 (12.7) | 64.6 (13.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 282 | 31 | 313
  Female | 155 | 49 | 204

OUTCOME MEASURES:

1. Primary Outcome: Rate of Non-recurrence at Week 52
Description: The non-recurrence rate (at 52 weeks) was determined by the endoscopy central review panel who were blinded to the investigator's assessment, based on the modified Los Angeles Classification using endoscopy photos were submitted by each of the institutions. Participants showing Grade A or above based on the modified Los Angeles Classification were included as a recurrence.
Time Frame: Week 52
Population: Central assessment Full Analysis Set (FAS) was defined as all randomized participants who received at least one dose of the study drug, and from whom the results of at least one endoscopic assessment was available. Data analysis excluded participants with missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily: Rabeprazole 10 mg or 20 mg were administered orally twice daily during the treatment period (unblinded), and 10 mg was administered once daily during the maintenance period (double-blind).
- Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily: Rabeprazole 10 mg or 20 mg were administered orally twice daily during the treatment period (unblinded), and 10 mg was administered twice daily during the maintenance period (double-blind).
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 163 | 161
Percentage of participants
  Non-recurrence | 44.8 [37.2 to 52.4] | 73.9 [67.1 to 80.7]
  Recurrence | 55.2 [NA to NA] — NA = not calculated | 26.1 [NA to NA] — NA = not calculated
Statistical Analysis 1: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Test type: Superiority or Other; p < 0.001, Chi-squared; P-value was calculated using chi-square test at two-sided significance level of alpha = 0.05

2. Secondary Outcome: Rate of Non-recurrence at Weeks 12 and 24
Description: The non-recurrence rate (up to 52 weeks) was determined by the endoscopy central review panel who were blinded to the investigator's assessment, based on the modified Los Angeles Classification using endoscopy photos were submitted by each of the institutions. Participants showing Grade A or above based on the modified Los Angeles Classification were included as a recurrence. The 95% CI was calculated by normal approximation.
Time Frame: Weeks 12 and 24
Population: Central assessment FAS. Data analysis excluded participants with missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 170 | 173
Percentage of participants
  Week 12, Non-recurrence: number analyzed (Participants) | 168 | 171
  Week 12, Non-recurrence | 62.5 [55.2 to 69.8] | 92.4 [88.4 to 96.4]
  Week 12, Recurrence: number analyzed (Participants) | 168 | 171
  Week 12, Recurrence | 37.5 [NA to NA] — NA = not calculated | 7.6 [NA to NA] — NA = not calculated
  Week 24, Non-recurrence: number analyzed (Participants) | 165 | 168
  Week 24, Non-recurrence | 55.8 [48.2 to 63.3] | 85.1 [79.7 to 90.5]
  Week 24, Recurrence: number analyzed (Participants) | 165 | 168
  Week 24, Recurrence | 44.2 [NA to NA] — NA = not calculated | 14.9 [NA to NA] — NA = not calculated
Statistical Analysis 1: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Comparison at Week 12; Test type: Superiority; p < 0.001, Chi-squared; P-value was calculated using chi-square test at a two-sided significance level of alpha = 0.05
Statistical Analysis 2: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Comparison at Week 24; Test type: Superiority; p < 0.001, Chi-squared; P-value was calculated using chi-square test at two-sided significance level of alpha = 0.05

3. Secondary Outcome: Cumulative Non-recurrence Rate at Week 52
Description: Non-recurrence rate at Week 52 was estimated using the Kaplan-Meier method.
Time Frame: Week 52
Population: Central assessment FAS
Measure: Number (95% Confidence Interval); unit: Percentage of non-recurrence
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 170 | 173
Percentage of non-recurrence | 41.5 [33.0 to 49.8] | 71.4 [62.8 to 78.4]
Statistical Analysis 1: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.23 to 0.49]

4. Secondary Outcome: Percentage of Participants With Heartburn (Daytime / Nighttime) During the Maintenance Therapy Period
Description: A comparison of the rabeprazole 10 mg once daily group and the rabeprazole 10 mg twice daily group was performed for participants who did not exhibit daytime or nighttime heartburn at Week 0 of the Maintenance Therapy Period. Heartburn is a burning sensation in the stomach or lower chest; it is worsened by bending or pressure on the abdomen. Heartburn frequency was rated from 0-day (no) to 7-day (always) and severity was graded on a 3-point scale (mild, moderate, severe). Heartburn was evaluated in the daytime (from wake-up time to time for bed) and nighttime (from time for bed to wake-up time).
Time Frame: From Week 4 up to Week 52
Population: Central assessment FAS - LOCF. Analysis was carried out on participants who were determined to be free of symptoms at maintenance therapy entry.
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 138 | 137
Percentage of participants
  Heartburn (yes) | 23.2 | 8.0
  Heartburn (no) | 76.8 | 92.0
Statistical Analysis 1: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Test type: Superiority; p < 0.001, Chi-squared; P-value was calculated using chi-square test at two-sided significance level of alpha = 0.05; Group difference = -15.2, 95% CI 2-sided [-23.5 to -6.8] — Group difference (percentage of participants) = Arm D (percentage of participants) - Arm C (percentage of participants) 95% CI was calculated based on normal approximation

5. Secondary Outcome: Frequency of Heartburn (Daytime / Nighttime) During the Maintenance Therapy Period
Description: A comparison of rabeprazole 10 mg once daily group and the rabeprazole 10 mg twice daily group shall be performed for participants who did not exhibit daytime or nighttime heartburn at 0 weeks of the maintenance therapy period. Daytime and nighttime heartburn, and nighttime sleep disorders shall likewise be compared. For the participants who had recurrence, values at the final evaluation were imputed using a last observation carried forward (LOCF) method.
Time Frame: From Week 4 up to Week 52
Population: Central assessment FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 170 | 173
Percentage of participants
  0 Days (no symptoms) | 85.2 | 85.1
  1 to 2 Days (occasional symptoms) | 12.3 | 11.2
  3 to 4 Days (sometimes had symptoms) | 1.9 | 0.6
  5 to 6 Days (often had symptoms) | 0.0 | 1.9
  7 Days (always had symptoms) | 0.6 | 1.2

6. Secondary Outcome: Severity of Heartburn (Daytime / Nighttime) During the Maintenance Therapy Period
Description: A comparison of the rabeprazole (10 mg once daily group) and the rabeprazole (10 mg twice daily group) was performed for participants who did not exhibit daytime or nighttime heartburn at Week 0 of the Maintenance Therapy Period. The presence or absence of heartburn was assessed by the investigators during medical interviews. The heartburn incidence during each of the 7-day periods immediately before visiting the hospital was assessed on a scale of five stages based on the number of days with symptoms: 0 (no symptoms), 1 to 2 (occasional symptoms), 3 to 4 (sometimes had symptoms), 5 to 6 (often had symptoms), and 7 (always had symptoms). The incidence was tabulated by an analysis classifying the states into two groups: "no symptom group" (0 days with symptoms) and "with symptoms group" (1 day or more with symptoms). The severity of heartburn was as below: Mild (feel heartburn but tolerable), Moderate (feel heartburn and hard), and Severe (feel heartburn and terrible).
Time Frame: From Week 4 up to Week 52
Population: Central assessment FAS - LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 170 | 173
Percentage of participants
  None | 85.2 | 85.1
  Mild | 14.8 | 14.3
  Moderate | 0.0 | 0.6
  Severe | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With Sleep Disorders During the Maintenance Therapy Period
Description: Sleep disorders were defined as the condition of lack of dead sleep and arousal during sleep arising from heartburn or acid reflux. Sleep disorders during each of the 7-day periods immediately before visiting the hospital were assessed. Evaluation of sleep disorders arising from heartburn or acid reflux included recording if sleep-inducing drugs were being taken before enrollment; their type, method of use, and dosage. It was requested that no changes in sleep-inducing drug be made after enrollment. Sleep disorders were rated from 0-day (no) to 7-day (always). The incidence of sleep disorder was tabulated by an analysis classifying the stages into two groups: "No" (0 days with sleep disorder) and "Yes" (1 or more days with sleep disorder). Heartburn was evaluated prior to 7 days of each visit.
Time Frame: From Week 4 up to Week 52
Population: Central assessment FAS. Participants who did not have sleep disorder due to nighttime heartburn or swallowing at the time of maintenance of the Maintenance Therapy Period, participants whose visit data was not missing.
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 157 | 158
Percentage of participants
  Sleep disorders from heartburn/acid reflux (yes) | 2.5 | 2.5
  Sleep disorders from heartburn/acid reflux (no) | 97.5 | 97.5
Statistical Analysis 1: Comparison: Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily vs Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily; Test type: Superiority; p = 0.992, Chi-squared — P-value was calculated using chi-square test at two-sided significance level of alpha = 0.05; Group difference = 0.0, 95% CI 2-sided [-3.5 to 3.5] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Frequency of Sleep Disorders During the Maintenance Therapy Period
Description: Sleep disorders were defined as the condition of lack of dead sleep and arousal during sleep arising from heartburn or acid reflux. Evaluation of sleep disorders arising from heartburn or acid reflux included recording if sleep-inducing drugs were being taken before enrollment; their type, method of use, and dosage. It was requested that no changes in sleep-inducing drug be made after enrollment. Sleep disorders were rated from 0-day (no) to 7-day (always). Heartburn was evaluated prior to 7 days of each visit.
Time Frame: From Week 4 up to Week 52
Population: Central assessment FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 170 | 173
Percentage of participants
  0 Day (none) | 96.9 | 98.1
  1 to 2 Days (occasional symptoms) | 2.5 | 0.6
  3 to 4 Days (sometimes had symptoms) | 0.6 | 0.0
  5 to 6 Days (often had symptoms) | 0.0 | 0.6
  7 Days (always had symptoms) | 0.0 | 0.6

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Safety was assessed by monitoring and recording all adverse events (AEs) and SAEs, regular monitoring of hematology, clinical chemistry, urine values, and regular measurement of vital signs. All AEs were graded on a 3-point scale; 1) mild was defined as discomfort that did not interfere with normal daily activities, 2) moderate was defined as discomfort that interfered with normal activities, and 3) severe was defined as discomfort that interfered with the ability to work or normal daily activities were impossible. SAEs were medical events that led to death, were life-threatening, required hospitalization or prolongation of hospitalization, caused persistent disability, or resulted in a congenital abnormality. TEAEs were AEs with an onset date on or after the first dose of study drug and up to 30 days after receiving the last dose of study drug. Treatment-related AEs were medical events that were considered by the investigator to be possibly or probably related to rabeprazole.
Time Frame: From date of first dose up to 30 days after the last dose of study drug, up to approximately 1 year 3 months (Treatment Period; 8 weeks, Maintenance Therapy Period; 52 weeks, and Follow-up Period; 30 days)
Population: Safety analysis set was the group of participants who received at least one dose of study drug (rabeprazole) in the Treatment Period or Maintenance Period and had at least one post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once daiArm C: Rabeprazole 10 mg or 20 mg were administered orally twice daily during the treatment period (unblinded), and 10 mg was administered once daily during the maintenance period (double-blind).
Arm/Group | Rabeprazole: 10 mg Twice Daily | Rabeprazole: 20 mg Twice Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once daiArm C | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
Number analyzed (Participants) | 437 | 80 | 178 | 181
Participants
  TEAEs | 111 | 21 | 111 | 125
  Treatment-related TEAEs | 20 | 1 | 7 | 11
  Severe TEAEs | 2 | 1 | 4 | 3
  Serious TEAEs | 6 | 4 | 11 | 17

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study drug, up to approximately 1 year 3 months (Treatment Period; 8 weeks, Maintenance Therapy Period; 52 weeks, and Follow-up Period; 30 days)
Description: Treatment-emergent adverse events and serious adverse events were reported. The safety analysis set was the group of participants who received at least one dose of study drug (rabeprazole) in the Treatment Period or Maintenance Therapy Period and had at least one post-dose safety assessment. All AEs were graded on a 3-point scale (mild, moderate, severe).
Arm/Group | Rabeprazole: 10 mg Twice Daily | Rabeprazole: 20 mg Twice Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/437 | 0/80 | 1/178 | 0/181
Serious Adverse Events (participants affected / at risk) | 6/437 | 4/80 | 11/178 | 17/181
Other Adverse Events (participants affected / at risk) | 63/437 | 12/80 | 75/178 | 87/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole: 10 mg Twice Daily (N=437) | Rabeprazole: 20 mg Twice Daily (N=80) | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily (N=178) | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily (N=181)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Drowning (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole: 10 mg Twice Daily (N=437) | Rabeprazole: 20 mg Twice Daily (N=80) | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Once Daily (N=178) | Rabeprazole: 10 or 20 mg Twice Daily, Then 10 mg Twice Daily (N=181)
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 3 | 10
Dental caries (Gastrointestinal disorders) | 0 | 1 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3 | 6
Constipation (Gastrointestinal disorders) | 3 | 1 | 4 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 5
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 4 | 1
Pyrexia (General disorders) | 2 | 1 | 1 | 4
Nasopharyngitis (Infections and infestations) | 25 | 5 | 32 | 33
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 9 | 10
Pharyngitis (Infections and infestations) | 4 | 0 | 5 | 8
Influenza (Infections and infestations) | 2 | 0 | 5 | 4
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 5
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 4 | 6
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 4 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Headache (Nervous system disorders) | 3 | 1 | 5 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 6 | 8
Hypertension (Vascular disorders) | 4 | 1 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other